CLINICAL TRIAL: NCT06897098
Title: Autologous Cartilage Implantation: Safety Study for Focal Chondral Lesions in the Knee and the Ankle : Open Cohort, Small Sample Size With 12 Months Follow-Up
Brief Title: Regeneration of Knee and Ankle Cartilage From Autologous Cartilage Mini-grafts (From the Patient's Own Cells)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanarix SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 701146; 701146 (CTI.02) (Other: Swissmedic); 2019-01727 (Other: BASEC); 52372 (Other: HumRes); 000004042 (Other: SNCTP)
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cartilage Repair
Keywords: Cartilage repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous Cartibeads (Experimental): Implantation of autologous cartilage mini-grafts (Cartibeads)
  Interventions: Biological: Implantation of autologous cartilage mini-grafts (Cartibeads)

INTERVENTIONS:
Biological: Implantation of autologous cartilage mini-grafts (Cartibeads) — 1. st surgery: cartilage biopsy harvest by minimally invasive surgery (arthroscopy or mini arthrotomy).
  2. nd surgery: Implantation of autologous cartilage mini-grafts (Cartibeads) by minimally invasive surgery (arthroscopy or mini arthrotomy). Cartibeads should entirely fill the defect zone, followed by a thin layer of surgical glue (TISSEEL Fibrin Sealant).

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of implanting autologous cartilage mini-grafts (or Cartibeads) into cartilage defects in the knee and ankle.

Cartibeads are engineered from autologous articular chondrocytes (from the patient's own cartilage cells). A small cartilage biopsy (~50 to 150 mg according to lesion size to be treated) is collected from a minimal weight bearing zone of the patient's articulation. Chondrocytes are extracted from the biopsy and expanded in culture. Our patented, standardized methodology then allows expanded cells to recover their capacity of producing hyaline matrix and to form cartilage mini-grafts (Cartibeads). These grafts are beads of 1 to 2 mm in diameter and have similar characteristics to native hyaline cartilage.

Autologous Cartibeads are implanted into the patient's cartilage defect. Patients are then followed for 12 months for assessment of study endpoints, with safety being the primary outcome.

ELIGIBILITY:
Key inclusion criteria:

* Cartilage focal lesion(s) ≥ 1.5 cm2 and ≤ 10 cm2
* ICRS grade 3 or 4
* Pain for 3 months or more
* Aged over 18 years

Key exclusion criteria

* Inability to undergo MRI
* Cartilage specific surgery within 12 months from baseline
* Cartilage therapeutic injection within 3 months from baseline
* Radiologically apparent degenerative joint disease (K&L grade >1)
* Chronic inflammatory arthritis and/or infectious arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-04-02 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
Safety | From enrolment to the end of follow-up at 12 months
  Recording, identifying, documenting and reporting all Serious Adverse Events (SAEs) and Adverse Events (AEs).

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - Center for Sports Medicine and Exercise, Hirslanden Clinique La Colline, Geneva, Canton of Geneva
  - Geneva University Hospitals (HUG), Geneva, Canton of Geneva
  - Ente Ospedaliero Cantonale (EOC), Lugano, Canton Ticino

IPD SHARING:
Plan to Share IPD: No